CLINICAL TRIAL: NCT07341139
Title: Is Long-Term Blood Storage Related With Increased Mortality and Adverse Effects in Severely Injured Trauma Patients?
Brief Title: Blood Storage Related Mortality and Adverse Effects in Trauma Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Kocaeli City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: AS-Blood
Record Dates: First submitted 2025-12-17; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Transfusion Adverse Reaction; Major Trauma; Blood Product Transfusion for All Conditions
Keywords: blood storage; Transfusion; Trauma; Red Blood Cell
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: The study will include patients aged 18-75, with an ISS >15, who presented directly from the injury scene and received massive transfusion (defined as >10 packed RBC (PRBC) units in the first 24 hours or ≥3 units in 1 hour) between January 1, 2023, and October 1, 2025. Data will be extracted from hospital information systems and anesthesia records. The storage duration for each transfused unit (from collection to transfusion) will be recorded.

SUMMARY:
The purpose of this retrospective study is to examine the following factors related to blood storage time in severely injured trauma patients who received large blood transfusions:

1. The effect of blood storage time on the patient's 28-day mortality rate.
2. The relationship between storage time and other health problems that the patient may develop (such as heart disease, vascular occlusion, respiratory failure, infection, and organ failure).

For this purpose, patients aged 18-75 who were admitted directly from the scene of injury and received large transfusions at Jacksonville Shands Hospital between January 1, 2023, and October 1, 2025, will be included. Data will be obtained from hospital information systems and anesthesia records

DETAILED DESCRIPTION:
Is Long-Term Blood Storage related with increased mortality and adverse effects in severely injured trauma patients?

Abstract

Background: Severe trauma remains a significant cause of mortality, often necessitating massive transfusion. During storage, red blood cells (RBCs) and whole blood units develop "storage lesions," encompassing biochemical and structural deteriorations such as oxidative damage to hemoglobin, metabolic derangements (e.g., lactate accumulation, adenosine triphosphate (ATP) and 2,3-diphosphoglycerate (2,3-DPG) depletion), and increased vesiculation. These changes are hypothesized to contribute to adverse clinical outcomes, including impaired microvascular perfusion, endothelial injury, hypercoagulability, inflammation, multi-organ dysfunction, and increased mortality. While numerous observational studies and meta-analyses suggest an association between prolonged blood storage duration and worse outcomes, large randomized controlled trials (RCTs) have yielded conflicting results. The impact of storage age on high-risk trauma patients requiring massive transfusion remains particularly uncertain.

Objective: This study aims to evaluate the effect of RBC and whole blood storage duration on 28-day mortality in severely injured trauma patients (Injury Severity Score (ISS) >15) undergoing massive transfusion. A secondary objective is to assess the relationship between storage duration and morbidity, including complications such as cardiac ischemia, thromboembolic events, acute respiratory failure, nosocomial infection, and multiple organ failure.

Methods: A single-center retrospective cohort study will be conducted at the University of Florida Jacksonville Shands Hospital. The study will include patients aged 18-75, with an ISS >15, who presented directly from the injury scene and received massive transfusion (defined as >10 packed RBC (PRBC) units in the first 24 hours or ≥3 units in 1 hour) between January 1, 2023, and October 1, 2025. Data will be extracted from hospital information systems and anesthesia records. The storage duration for each transfused unit (from collection to transfusion) will be recorded. Blood products are preserved with Adsol AS-1 additive solution, allowing storage of packed RBCs for 42 days and whole blood for 21 days.

Patients will be analyzed based on the product type (PRBCs vs. whole blood) and stratified into storage duration groups: Group 1 (0-7 days), Group 2 (8-14 days), Group 3 (15-21 days), and Group 4 (≥22 days, for PRBCs only). Comprehensive data will be collected, including demographics, injury mechanism, physiological parameters (vital signs, blood gas analyses including lactate, HCO₃, Hb, pH), laboratory values (e.g., creatinine), transfusion volumes (RBC, fresh frozen plasma (FFP), platelets, cryoprecipitate), fluid administration, urine output, vasopressor requirements, and perioperative complications. Outcomes of interest are 28-day mortality, morbidity endpoints, and lengths of intensive care unit (ICU) and hospital stay.

Statistical Analysis: Statistical analyses will be performed using R software. Descriptive statistics will summarize the data. Normality will be assessed using the Shapiro-Wilk test. Group comparisons will utilize t-tests, Mann-Whitney U tests, ANOVA, or Wilcoxon tests as appropriate. Categorical data will be compared using Pearson's chi-square or Fisher's exact tests. Correlations will be assessed via Spearman's analysis. Linear and logistic regression models will identify factors influencing continuous outcomes (e.g., ICU stay) and binary outcomes (e.g., mortality, complications), respectively. Survival analysis will employ Kaplan-Meier curves and the Log-Rank test. A p-value <0.05 will be considered statistically significant.

Conclusion: This retrospective cohort study seeks to clarify the contentious relationship between the age of transfused blood and clinical outcomes in a high-risk population of major trauma patients requiring massive transfusion. By specifically focusing on this vulnerable group and employing detailed stratification of storage duration, the study aims to provide evidence on whether the transfusion of older blood units is associated with increased 28-day mortality and higher morbidity. The findings could inform blood bank inventory management and transfusion practices in trauma resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-75 years of age,
* Injury Severity Score>15 and have received massive blood transfusions in our hospital from 1 January 2015 to 31 December 2025
* The patients admitted because of trauma and undergoing surgery

Exclusion Criteria:

* Patients with known cardiac or vascular diseases such as heart failure or malignant hypertension, those under anticoagulant treatment
* Patients with known serious kidney (on dialysis), lung, liver diseases, those under anticoagulant treatment
* Super obese patients with body mass index (BMI) 50 or above

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In our study, patients between the ages of 18-75, directly from the scene of injury, ISS>15 and who received massive blood transfusion (>10 packed RBC units in the first 24 hours, with an alternative definition of greater than or equal to 3 packed RBC units transfused in 1 hour) will be included in the study at University of Florida Jacksonville Shands Hospital between the dates 1 January 2023 to 1 31 December 2025.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
28-day Mortality | At the day of 28 after massive blood transfusion
  The aim of this study was to evaluate the effect of red blood cell and whole blood storage duration on 28-day mortality in severely injured trauma patients (injury severity score >15) undergoing massive transfusion.

SECONDARY OUTCOMES:
28-day Morbidity | At the day of 28 after massive blood transfusion
  On the 28th day after the blood transfusion, patients will be assessed for morbidities including complications such as cardiac ischemia, thromboembolic events, acute respiratory failure, nosocomial infection, and multiple organ failure.

CONTACTS AND LOCATIONS:
Overall Officials: ayten saracoglu, Principal Investigator — University of Florida
Locations (1):
- UF Health Jacksonville (Shands Hospital), Jacksonville, Florida, United States